CLINICAL TRIAL: NCT01618344
Title: Use of a Smart-phone Medication Reminder Application to Promote Adherence to Oral Medications by Adolescents and Young Adults(AYA) With Cancer
Brief Title: Smart-phone Application to Promote Medication Adherence in Adolescents and Young Adults (AYA) With Cancer
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Yelena Wu, Principal Investigator, University of Utah
Other Study IDs: SCH-13929
Record Dates: First submitted 2012-04-25; First posted 2012-06-13 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Neoplasms
Keywords: neoplasms; adolescent; young adult; medication adherence
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To explore use of a smart-phone medication reminder application to promote adherence to oral medications by AYA with cancer.

DETAILED DESCRIPTION:
Non-adherence to oral medications is a prevalent problem in adolescents and young adults (AYA) with cancer that may impact both survival and quality of life while on treatment. The purpose of this study is to explore use of a smart-phone medication reminder application to promote adherence to oral medications by AYA with cancer. The study's primary aim is to explore the feasibility and acceptability of using a smart-phone medication reminder application to promote adherence to oral medications by AYA with cancer as well as to characterize application use. Secondary aims include: 1) to obtain initial estimates of intervention effect- measured by pre-intervention to post-intervention differences in perceived behavioral control for adherence, intention to adhere, and adherence behavior - to inform design of a future trial powered to detect a clinically significant effect of smart-phone medication reminder application use on adherence to oral medications; and 2) to examine the relationships among perceived behavioral control for adherence, intention to adhere, and adherence behavior. A pre-post single group design will be used. Data will be collected weekly for 4 weeks before introduction of the intervention and for 8 weeks following introduction of the intervention. Analytic approaches will include descriptive statistics and generalized estimating equation (GEE) modeling.

ELIGIBILITY:
Inclusion criteria:

1)15-29 year olds receiving treatment for any type of cancer, either primary or recurrent/relapsed disease.

2) Patient has completed at least one month of therapy

3)Patient is expected to remain on therapy for 3 month duration of study

4) Patient has an iPhone, iPad, or iTouch running iOS 4.0 or later

5) Patient is willing to use a smart-phone medication reminder application-

Exclusion Criteria:

1)Patients who are unable to speak/read/write English as required for use of smart-phone medication reminder application and completion of study measures.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinics for patients be treated for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PhD, Principal Investigator — Huntsman Cancer Institute; Lauri Linder, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Smart-phone Medication Reminder Application: All participants were provided with the medication reminder application, and were instructed on how to program the application based on their individual medication dosing schedules. At the scheduled times, the application prompted participants to take their medications.
Period: Overall Study
Arm/Group | Smart-phone Medication Reminder Application
Started | 32
Completed | 23
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Participants: All participants
Arm/Group | Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Acceptability of Using a Smart-phone Medication Reminder Application to Promote Adherence to Oral Medications by AYA With Cancer.
Description: Feasibility was assessed through participants' application usage and responses to self-reported questions about their use of the application. Acceptability was assessed through participants' perceived ease of use and perceived usefulness of the application.
Time Frame: ongoing study weeks 5-12
Measure: Count of Participants; unit: Participants
Arm/Group | Participants
Number analyzed (Participants) | 23
Participants
  Used application at least once | 21
  Took medication immediately upon getting reminder | 13

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months per participant.
Description: Any adverse events would have been reported to the University of Utah Institutional Review Board via a report form.
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
Small pilot trial (single group). Pre-post measurements only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT01618344/Prot_SAP_000.pdf